CLINICAL TRIAL: NCT07125378
Title: Living Independence Through Functional Training (LIFT): Feasibility of Hybrid Task-Oriented Resistance Exercise Following Home Health Discharge
Brief Title: Living Independence Through Functional Training
Acronym: LIFT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202500835
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mobility Limitation; Cognitive Impairment
Keywords: Home-based intervention; Exercise; Older adults; Activities of daily living; Mobility; Cognition
MeSH Terms: conditions — Mobility Limitation; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Intervention Model Description: One group with repeated measures at baseline, post-intervention, and one-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LIFT (Experimental): Participants will receive a task-oriented resistance exercise program at home.
  Interventions: Behavioral: Task-oriented resistance exercise

INTERVENTIONS:
Behavioral: Task-oriented resistance exercise — The intervention program includes progressive resistance exercise and daily activity exercise, delivered over a six-week period with an ideal frequency of three sessions per week. Progressive resistance exercise will be provided through a combination of in-person and online sessions, while daily activity exercise will be delivered exclusively in person.

SUMMARY:
The purpose of the research is to evaluate the feasibility and benefits of a six-week hybrid task-oriented resistance exercise program for older adults who have been recently discharged from home health care.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 65 and 90 years
* community-dwelling
* live within a 50-mile radius of the study site with wireless connectivity in the area
* mobility limitations as indicated by self-reported of using a mobility aid or having unsteady gait or walking slower than before
* cognitive decline as indicated by a score < 12 on Mini MoCA Version 2.1
* a care partner or adult family member living in the home or nearby
* willing to wear an activity tracker during the study period

Exclusion Criteria:

* plan to receive skilled rehabilitation services
* plan to move away outside the study area in two months
* reside in an assisted living or long-term care facility or plan to relocate to such a facility in the next three months
* severe vision or hearing loss that impedes activity performance or communication
* unable to stand or walk even with a mobility aid
* unable to follow a one-step command or carry on a conversation over the phone
* unable to commit to the six-week exercise program
* contradictions to resistance exercise, such as the end-stage heart failure
* a terminal disease or on hospice care
* a neurological condition affecting motor skills
* not able to provide consent.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Baseline, 8 weeks, and 12 weeks.
  The score ranges from 0 to 12, with a score of 12 indicating the best physical functioning of the lower extremity.
Montreal Cognitive Assessment | Baseline, 8 weeks, and 12 weeks.
  The score ranges from 0 to 30, with a score of 30 indicating the best global cognitive function.

SECONDARY OUTCOMES:
Timed Up and Go Test-Single Task. | Baseline, 8 weeks, and 12 weeks.
  Time in seconds to complete the test, with a longer time indicating poor functional mobility.
Timed Up and Go-Dual Task | Baseline, 8 weeks, and 12 weeks.
  Time in seconds to complete the task, a longer time indicating the interference of the dual task effect on mobility.
List Sorting Working Memory Test | Baseline, 8 weeks, and 12 weeks.
  The raw score ranges from 0 to 24, with a higher score indicating better working memory. The raw score is converted to a Change Sensitive Score.
Dimensional Change Card Sort Test | Baseline, 8 weeks, 12 weeks.
  The raw score ranges from 0 to 30, with a higher score indicating better executive function. The raw score is converted to a Change Sensitive Score.
Flanker Inhibitory Control and Attention Test | Baseline, 8 weeks, and 12 weeks
  The raw score ranges from 0 to 30, with a higher score indicating better executive function and attention. The raw score is converted to a Change Sensitive Score.
Pattern Comparison Processing Speed Test | Baseline, 8 weeks, and 12 weeks
  The raw score ranges from 0-133, with a higher score indicating better processing speed. The raw score is converted to a Change Sensitive Score.
Speeded Matching Test | Baseline, 8 weeks, 12 weeks
  The score ranges from 0 to 130, with a higher score indicating better speed of processing. The raw score is converted to a Change Sensitive Score.
Oral Symbol Digit Test | Baseline, 8 weeks, and 12 weeks
  The raw score ranges from 0 to 143, with a higher score indicating better processing speed. The raw score is converted to a Rasch score.

OTHER OUTCOMES:
Patient Health Questionnaire-9 | Baseline, 8 weeks, 12 weeks.
  The score ranges from 0 to 27, with a higher score indicating a higher degree of depression.
Pain, Enjoyment of Life and General Activity Scale | Baseline, 8 weeks, and 12 weeks.
  The score ranges from 0 to 10, with a higher score indicating greater pain and interference with life by pain.
Activity Measure for Post-Acute Care to measure everyday activity performance | Baseline, 8 weeks, and 12 weeks.
  The score ranges from 0 to 71, with a higher score indicating better mobility, daily activity function, or daily cognitive ability.
Step counts | From enrollment to the end of intervention at 8 weeks.
  The number of step counts, a higher number indicates a higher level of physical activity.
Sleep efficiently | From enrollment to the end of the intervention at 8 weeks.
  A ratio score of total sleep time divided by total time in bed per night, ranging from 0 to 1. A higher score indicates better sleep quality.
Program satisfaction | 8 weeks
  A score ranges from 0 to 6, with a higher score indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chiung-ju Liu Associate Professor, phD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - College of Public Health and Health Professions, University of Florida, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie the results in a publication
Time Frame: Data requests can be submitted starting 3 months after article publication, and the data will be made accessible for up to 12 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and able to provide a research proposal and data usage agreement. Please contact the trial principal investigator.